CLINICAL TRIAL: NCT05070468
Title: The Effect of Using Dexamethasone Tablets Vaginally On Improving Cervical Bishop Score in Nulliparous Pregnant Women. A Randomized Clinical Trial
Brief Title: Effect of Dexamethasone on Labor Induction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alborz Medical University (Other Government)
Responsible Party: Principal Investigator, Matineh Nirouei, Principal Investigator, Alborz Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.ABZUMS.REC.1399.067
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Dexamethasone; Pregnancy
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Subjects are assigned to two groups by randomization block balanced method allocation and using quadruple blocks. In this case, there are 6 modes And in each case, 2 people will be in the control group and 2 people will be in the intervention group. Thus, by using the table of random numbers and assigning the numbers 1 to 6 to groups of 4 people, people are finally assigned to two groups of intervention and control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pregnant women with a gestational age of 38 weeks and older admitted to Labor Of Kamali Hospital, for termination of pregnancy, by accident and based on the coding done by a statistician to identify groups of users of pill A or pill B, 14 pills are used vaginally . The client and the researcher are blinded and the pharmacist delivers the dexamethasone and placebo tablets with codes A and B to the researcher.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Prescribing Vaginally Dexamethasone tablets to the Group A
  Interventions: Drug: Dexamethasone 0.5mg
- Group B (Placebo Comparator): Prescribing Vaginally placebo tablets to the Group B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone 0.5mg — Pregnant women with a gestational age of 38 weeks and older admitted to Labor Of Kamali Hospital, for termination of pregnancy, by accident and based on the coding done by a statistician to identify groups of users of pill A or pill B, 14 pills are used vaginally . The client and the researcher are blinded and the pharmacist delivers the dexamethasone and placebo tablets with codes A and B to the researcher.
  Other Names: Pill A
  Arms: Group A
Drug: Placebo — Pregnant women with a gestational age of 38 weeks and older admitted to Labor Of Kamali Hospital, for termination of pregnancy, by accident and based on the coding done by a statistician to identify groups of users of pill A or pill B, 14 pills are used vaginally . The client and the researcher are blinded and the pharmacist delivers the dexamethasone and placebo tablets with codes A and B to the researcher.
  Other Names: Pill B
  Arms: Group B

SUMMARY:
Pregnant women with a gestational age of 38 weeks and older admitted to Labor Of Kamali Hospital, for termination of pregnancy, by accident and based on the a statistician did coding to identify groups of users of pill A or pill B, 14 pills are used vaginally. The patients and the researcher is blinded and the pharmacist delivers the dexamethasone and placebo tablets with codes A and B to the researcher.

DETAILED DESCRIPTION:
Study design:

This study was a clinical trial with the control group, blinded, randomized with a block method that was done at Kamali Hospital, Karaj, Iran.

This study was carried out between October 2019 and June 2021. At first, the researchers registered this study on the RCT(randomized controlled trial) site with the following number: IR.ABZUMS.REC1399.067.

A written consent form was obtained from all patients and the ethics committee of Alborz University of Medical Sciences confirmed the study protocol.

Study selection:

The sample size required to compare the mean of the two groups, with a 95% confidence interval and 90% test power, and considering the technical difference of 0.5 hours, was estimated to be 84 people. Then patients, randomly assigned using the block method with statistician help, were divided into two groups of 42 cases and control.

The present study was performed on 82 full-term pregnant females (38 weeks or more).they had an indication for termination of pregnancy, by accident, and based on the coding done by a statistician to identify groups of users of pill A or pill B, 14 pills are used vaginally. The client and the researcher are blinded and the pharmacist delivers the dexamethasone and placebo tablets with codes A and B to the researcher. Group A received 14 dexamethasone tablets with a dose of 0.5 mg for vaginal use and also group B received 14 placebo tablets for vaginal use.

Patients who were Iranian, Prim gravid pregnancy with Normal Body Mass Index (BMI), Single Pregnancy presentation cephalic in Sonography, Aged 18 years old to 35 years old, Gestational age 38 weeks, Bishop score 2 and less, with Normal Non-Stress Test (NST), Estimate of Fetus Weight 2500-4000 gr and didn't take hormonal, herbal and chemical drugs and having a healthy water bag were enrolled to this Study.

Patients who had Medicine and Midwifery Complications, Lack of Desire for Cooperation, Fetal Immobility, and Maternal Bleeding were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Iranian Women
* Primigravid pregnancy
* Normal of Body Mass Index
* Single Pregnancy
* presentation cephalic in sonography
* Gestational age 38 weeks
* Bishop score 2 and less
* Normal Non Stress
* Test Estimate of Fetus Weight 2500-4000 gr
* Didn't take hormonal, herbal and chemical drugs
* having a healthy water bag

Exclusion Criteria:

* Have Medicine And Midwifery Complication
* Lack of Desire for Cooperation
* Fetal Immobility
* Maternal Bleeding

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masoumeh Farahani, Doctor, Study Director — Assistant Professor of Alborz University of Medical Sciences
Locations (1):
- Alborz university of medical sciences, Karaj, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farahani M, Nirouei M, Moghadam S, Hashemnejad M, Mashak B, Alinia T, Torabi S. The Effect of Using Dexamethasone Tablets Vaginally for Improving Cervical Bishop Score in Nulliparous Pregnant Women: A Randomized Clinical Trial. Curr Ther Res Clin Exp. 2023 Apr 6;98:100702. doi: 10.1016/j.curtheres.2023.100702. eCollection 2023. PMID 37101983

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone: Prescribing Vaginally Dexamethasone tablets to the Group A
  Dexamethasone 0.5mg: Pregnant women with a gestational age of 38 weeks and older admitted to Labor Of Kamali Hospital, for termination of pregnancy, by accident and based on the coding done by a statistician to identify groups of users of pill A or pill B, 14 pills are used vaginally . The client and the researcher are blinded and the pharmacist delivers the dexamethasone and placebo tablets with codes A and B to the researcher.
- Placebo: Prescribing Vaginally placebo tablets to the Group B
  Placebo: Pregnant women with a gestational age of 38 weeks and older admitted to Labor Of Kamali Hospital, for termination of pregnancy, by accident and based on the coding done by a statistician to identify groups of users of pill A or pill B, 14 pills are used vaginally . The client and the researcher are blinded and the pharmacist delivers the dexamethasone and placebo tablets with codes A and B to the researcher.
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 42 | 42
Completed | 41 | 42
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [22 to 31] | 23 [21 to 28.25] | 24 [22 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Count of Participants; unit: Participants]
  Illiterate | 4 | 6 | 10
  Primary school | 2 | 5 | 7
  Junior school | 14 | 7 | 21
  High school | 16 | 19 | 35
  Associate's degree | 2 | 2 | 4
  Bachelor's degree or higher | 4 | 3 | 7
Job [Count of Participants; unit: Participants]
  Unemployed | 37 | 40 | 77
  employed | 5 | 2 | 7
Gravidity and parity [Count of Participants; unit: Participants] — Gravidity (G) is the number of times a patient has been pregnant. This includes a current pregnancy. Parity (para) is the number of times a patient has given birth to a viable child. Abortion (ab) is the term used to describe a pregnancy that ended for any given reason, including both abortions and miscarriages.
  Participants
    G1ab1 | 42 | 40 | 82
    G1ab2 | 0 | 1 | 1
    G1ab3 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: First Bishop Score
Description: The total Bishop score is calculated by assessing the following five components of manual vaginal examination by a trained professional: Cervical dilation, Cervical effacement, Cervical consistency, Cervical position, and Fetal station.
  Dilation (score): closed(0), 1-2 cm (1), 3-4cm (2), 5>= (3) Effacement (score): 0-30% (0), 40-50% (1), 60-70% (2), 80%>= (3) Consistency (score): Firm (0), moderately firm (1), soft (2) Position (score): posterior (0), mid posterior (1), anterior(2) Station (score): -3 (0), -2 (1), -1 and 0 (2), +1 and +2 (3) The total Bishop's score which sums up all subscores can range from zero to 13, with zero meaning that the patient is not ready for induction and 13 indicating a better chance for successful induction for delivery (outcome).
Time Frame: at the beginning of the study
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 41 | 42
score on a scale | 1 [1 to 2] | 1 [1 to 2]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.618, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Second Bishop Score
Description: as for outcome 1
Time Frame: 6 hours after vaginally tablets installment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 41 | 42
score on a scale | 3.5 [2 to 4] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.483, Wilcoxon (Mann-Whitney)

3. Primary Outcome: The Latent Phase of Labor
Description: measured by Vaginal Examination
Time Frame: from the beginning of the study to the time of 6 cm dilation of cervix
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 41 | 42
hour | 4 [0 to 9] | 5 [0 to 8]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.571, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 20 hours
Groups:
- Group A; Group B: No deaths were recorded in the study, and no Serious Adverse Events were recorded in the study.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05070468/Prot_SAP_000.pdf